CLINICAL TRIAL: NCT00786474
Title: Bridging Anticoagulation in Patients Who Require Temporary Interruption of Warfarin Therapy for an Elective Invasive Procedure or Surgery
Brief Title: Effectiveness of Bridging Anticoagulation for Surgery (The BRIDGE Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00017344; 1U01HL086755-01A1 (NIH); 1U01HL087229 (NIH)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-01

CONDITIONS: Arterial Thromboembolic Events; Atrial Fibrillation
Keywords: Bridging Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dalteparin (Experimental)
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Placebo — Normal saline solution, dosage determined by weight, self-administered by patient twice a day
  Arms: Placebo
Drug: Dalteparin — Low molecular weight heparin (LMWH), dosage determined by weight, self-administered by patient twice a day
  Other Names: Fragmin
  Arms: Dalteparin

SUMMARY:
Blood thinners, such as warfarin, prevent blood clots from forming, thereby reducing the risk of a stroke or heart attack. When people undergo surgery or certain procedures, they must stop using warfarin to prevent too much bleeding during and after the surgery or procedure. Some doctors prescribe a different blood thinner, one that works more quickly and wears off more quickly, to bridge the gap between starting and stopping warfarin. However, this short-term treatment is expensive, may increase the risk of bleeding, and has not been proven effective. This study will determine whether a bridging blood thinner called dalteparin is helpful or harmful for people with atrial fibrillation who stop taking warfarin in preparation for surgery or a procedure.

DETAILED DESCRIPTION:
Approximately 2 million people in North America take the anticoagulant warfarin to prevent stroke, heart attack, and other events related to blood clots. Warfarin needs to be stopped before a person undergoes surgery or certain procedures because it can cause dangerous amounts of bleeding during and after surgery. Some doctors give a low molecular weight heparin (LMWH) to patients during the 2-week period when participants are without the effects of warfarin. The LMWH has the same effect as warfarin, but it acts and then leaves the system more quickly than warfarin. However, the LMWH is expensive, may increase the risk of bleeding, and has not been proven effective. This study will determine the safety and efficacy of an LMWH in adults with atrial fibrillation who stop warfarin in preparation for surgery.

Participation in this study will last between 36 and 67 days. Participation will involve nine points of contact with researchers, at least two of which will be in-person visits at the research clinic. The others will be conducted by phone. All points of contact will include assessments on possible bleeding and any new symptoms. The first two of these points of contact, will take place at the signing of the informed consent, which will involve a screening of medical records and random assignment of participants to receive either the LMWH dalteparin or placebo. Participants will self-administer a subcutaneous injection of their assigned treatment twice a day for 3 days before the surgery or procedure and for 6 days after. During the course of the study, when participants visit their primary physicians for regularly scheduled appointments, it will be recommended that they undergo two international normalized ratio (INR) tests of blood clotting ability between day 2 and 10 after the surgery or procedure. The remaining seven points of contact will occur sometime between the day before surgery and 37 days after surgery. One of the in-person visits will occur within the first week after surgery and will include assessments on possible bleeding, any new symptoms, and INR results.

ELIGIBILITY:
Inclusion Criteria:

* Receiving warfarin therapy for at least 3 months, administered to achieve an international normalized ratio (INR) range of 2.0 to 3.0
* Requiring temporary interruption of warfarin for pre-specified elective procedure or surgery
* Presence of one of the following conditions:

  1. Chronic (permanent or paroxysmal) nonvalvular atrial fibrillation, confirmed by at least one prior electrocardiography recording or pacemaker or acid citrate dextrose (ACD) interrogation
  2. Chronic (permanent or paroxysmal) valvular atrial fibrillation with evidence of mitral valvular heart disease, confirmed by the same criteria as nonvalvular atrial fibrillation
* Presence of at least one of the following major stroke risk factors:

  1. Older than 75 years of age
  2. Hypertension
  3. Diabetes mellitus
  4. Congestive heart failure or left ventricular dysfunction
  5. Previous ischemic stroke, systemic embolism, or transient ischemic attack (TIA)

Exclusion Criteria:

* Any mechanical prosthetic heart valve
* Stroke (ischemic or hemorrhagic), systemic embolism, or TIA within the past 12 weeks
* Venous thromboembolism (deep vein thrombosis and/or pulmonary embolism) within past 12 weeks
* Major bleeding within the past 6 weeks
* Severe renal insufficiency, measured through a calculated creatinine clearance of less than 30 mL/min
* Thrombocytopenia
* Life expectancy less than 1 month
* Condition that impairs compliance with trial protocol, such as cognitive impairment, an uncontrolled psychiatric condition, or geographic inaccessibility
* Pregnancy
* Allergy to heparin or history of heparin-induced thrombocytopenia
* Having one of the following surgeries or procedures during warfarin interruption:

  1. Cardiac surgery, such as coronary artery bypass or heart valve replacement
  2. Neurosurgery that is intracranial or intraspinal, such as tumor resection or aneurysm repair
  3. High-risk non-surgical procedures, such as brain biopsy
* Other surgical or non-surgical procedure that, at the discretion of the surgeon, precludes administration of therapeutic-dose low molecular weight heparin (LMWH) at any time in the post-procedure period
* More than one surgery planned during the trial period
* Prior participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1884 (Actual)
Dates: Start 2009-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Ortel, MD, Principal Investigator — Duke University; Victor Hasselblad, PhD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Wight JM, Columb MO. Perioperative bridging anticoagulation for atrial fibrillation-the first randomised controlled trial. Perioper Med (Lond). 2016 Jun 7;5:14. doi: 10.1186/s13741-016-0040-5. eCollection 2016. PMID 27280017
- [Derived] Douketis JD, Spyropoulos AC, Kaatz S, Becker RC, Caprini JA, Dunn AS, Garcia DA, Jacobson A, Jaffer AK, Kong DF, Schulman S, Turpie AG, Hasselblad V, Ortel TL; BRIDGE Investigators. Perioperative Bridging Anticoagulation in Patients with Atrial Fibrillation. N Engl J Med. 2015 Aug 27;373(9):823-33. doi: 10.1056/NEJMoa1501035. Epub 2015 Jun 22. PMID 26095867
- [Derived] Assaad B, Sesi VK, Figari R, Schultz L, Thummala N, Rehman M, Chandok A, Silverman A, Silver B. Antithrombotic management of stroke patients before colonoscopy. J Stroke Cerebrovasc Dis. 2013 Aug;22(6):733-6. doi: 10.1016/j.jstrokecerebrovasdis.2011.12.006. Epub 2012 Jan 12. PMID 22244711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6585 subjects were screened. 4701 were excluded, 1884 subjects enrolled and underwent randomization.
Period: Overall Study
Arm/Group | Placebo | Dalteparin
Started | 950 | 934
Completed | 913 | 891
Not Completed | 37 | 43
Not completed — Death | 5 | 4
Not completed — Withdrawal by Subject | 23 | 31
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dalteparin | Total
Number analyzed (Participants) | 950 | 934 | 1884
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (8.74) | 71.6 (8.88) | 71.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 248 | 502
  Male | 696 | 686 | 1382
Race/Ethnicity, Customized [Number; unit: participants]
  White | 860 | 849 | 1709
  Nonwhite | 88 | 82 | 170
  Unknown | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Arterial Thromboembolic Events
Description: The events are defined as arterial thromboembolism: stokes, transient ischemic attack and systemic embolism events were independently and blindly adjudicated
Time Frame: from subject signing of the consent until completed the study (Day -30 to Day +37)
Population: Of the 1,884 subjects enrolled in the trial, 71 discontinued participation and did not provide outcome data.
Measure: Number; unit: Arterial thromboembolic events
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 918 | 895
Arterial thromboembolic events
  Stroke | 2 | 3
  Transient Ischemic Attack | 2 | 0
  Systemic embolism | 0 | 0

2. Primary Outcome: Major Bleeding
Description: Major bleeding is defined as symptomatic bleeding associated with transfusion of more than two units of packed red blood cells or whole blood, or death
Time Frame: from subject signing of the consent until completed the study (Day -30 to Day +37)
Population: Of the 1,884 subjects enrolled in the trial, 71 discontinued participation and did not provide outcome data.
Measure: Number; unit: participants
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 918 | 895
participants | 12 | 29

3. Secondary Outcome: Number of Subjects With Death, Acute Myocardial Infarction, Deep Vein Thrombosis, or Pulmonary Embolism
Time Frame: from subject signing of the consent until completed the study (Day -30 to Day +37)
Population: Of the 1,884 subjects enrolled in the trial, 71 discontinued participation and did not provide outcome data.
Measure: Number; unit: participants
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 918 | 895
participants
  Death | 5 | 4
  Myocardial infarction | 7 | 14
  Deep-vein thrombosis | 0 | 1
  pulmonary embolism | 0 | 1

4. Secondary Outcome: Number of Participants With Minor Bleeding
Description: Minor bleeding is defined as symptomatic or clinically-overt bleeding that does not satisfy the criteria for major bleeding
Time Frame: from subject signing of the consent until completed the study (Day -30 to Day +37)
Population: Of the 1,884 subjects enrolled in the trial, 71 discontinued participation and did not provide outcome data
Measure: Number; unit: participants
Arm/Group | Placebo | Dalteparin
Number analyzed (Participants) | 918 | 895
participants | 110 | 187

ADVERSE EVENTS:
Time Frame: from subject signing of the consent until completed the study from Day -30 to Day +37
Description: Study only collected and reported serious adverse events
Arm/Group | Placebo | Dalteparin
Serious Adverse Events (participants affected / at risk) | 66/950 | 133/934
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=950) | Dalteparin (N=934)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Hypocoagulable State (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 3
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 3
Atrial Flutter (Cardiac disorders) | 1 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 4 | 5
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 2
Adrenal Haemorrhage (Endocrine disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric Perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Pancreatic Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 6
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cardiac Death (General disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholangitis (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Gallbladder Fistula (Hepatobiliary disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Arthritis Bacterial (Hepatobiliary disorders) | 0 | 1
Arthritis Infective (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Perirectal Abscess (Infections and infestations) | 0 | 1
Peritonsillar Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 5
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 5
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 3 | 4
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 | 0
Vaginal Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood Culture Positive (Investigations) | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperosmolar State (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient Ischaemic Attack (Nervous system disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 5
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Urethral Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Bladder Rupture (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No